CLINICAL TRIAL: NCT01721135
Title: A Randomised, Placebo Controlled, Four-way Cross-over Study to Assess Cardiac Re-polarisation Following Repeat Dosing With GSK2190915 and Placebo for Five Days, With Moxifloxacin as a Positive Control, in Healthy Male and Female Subjects.
Brief Title: A Study to Evaluate the Effect of Two Different Repeat Doses of GSK2190915 on the QTc Interval.
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was terminated due to toxicology findings after screening started but before first subject first dose.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 112360
Record Dates: First submitted 2012-11-01; First posted 2012-11-05 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Asthma
Keywords: moxifloxacin; GSK2190915; pharmacokinetics; QTc
MeSH Terms: conditions — Asthma | interventions — 3-(3-tert-butylsulfanyl-1-(4-(6-ethoxypyridin-3-yl)benzyl)-5-(5-methylpyridin-2-ylmethoxy)-1H-indol-2-yl)-2,2-dimethylpropionic acid; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- GSK2190915 100mg (Experimental): GSK2190915 100mg on days 1-5; moxifloxacin placebo on day 5
  Interventions: Drug: GSK2190915 100mg; Drug: moxifloxacin placebo; Drug: GSK2190915 placebo
- GSK2190915 1000mg (Experimental): GSK2190915 1000mg on days 1-5; moxifloxacin placebo on day 5
  Interventions: Drug: GSK2190915 200mg; Drug: moxifloxacin placebo
- moxifloxacin 400mg (Active Comparator): placebo tablet on days 1-5; moxifloxacin 400mg on day 5
  Interventions: Drug: moxifloxacin 400mg; Drug: GSK2190915 placebo
- placebo (Placebo Comparator): placebo tablet on days 1-5; moxifloxacin placebo on day 5
  Interventions: Drug: moxifloxacin placebo; Drug: GSK2190915 placebo

INTERVENTIONS:
Drug: GSK2190915 100mg — Film coated oral tablet
  Arms: GSK2190915 100mg
Drug: GSK2190915 200mg — Film coated oral tablet
  Arms: GSK2190915 1000mg
Drug: moxifloxacin 400mg — Film coated oral tablet
  Arms: moxifloxacin 400mg
Drug: moxifloxacin placebo — Film coated oral tablet
  Arms: GSK2190915 1000mg; GSK2190915 100mg; placebo
Drug: GSK2190915 placebo — Film coated oral tablet
  Arms: GSK2190915 100mg; moxifloxacin 400mg; placebo

SUMMARY:
This study is a randomized, placebo controlled, four way crossover, in which the the effect of GSK2190915 on the QTc interval is assessed. Healthy subjects will recieve a 5 day course of each of the following; oral placebo, GSK2190915 100mg, GSK2190915 1000mg and moxifloxacin 400mg (single dose) with a weeks washout prior to starting the next course. Key assessments include a 12- lead electrocardiogram and pharmacokinetic testing. Safety will be assessed by blood pressure, heart rate, clinical laboratory safety tests and collection of adverse events .

DETAILED DESCRIPTION:
This is a randomized, placebo controlled, four way crossover thorough QT study to evaluate the effect of repeat dose GSK2190915 on the QTc interval in healthy male and female subjects. Approximately 48 subjects will receive oral placebo, GSK2190915 (100mg or 1000mg) and moxifloxacin (400mg). GSK2190915 or matching placebo will be given once daily for 5 days with a moxifloxacin matching placebo given on Day 5. Moxifloxacin (positive control) will be given as a single-blind single dose on Day 5 with placebo administered on Days 1-4. Individual time-matched changes from baseline in QTcF (difference from placebo) for GSK2190915 will be determined 0-24 hours after dosing on Day 5 (primary endpoint). Secondary endpoints will include changes from baseline in QTcF, QTcB and QT interval at each timepoint after 5 days dosing of GSK2190915 and single dose moxifloxacin (400mg). Plasma concentrations on Day 5 (0-24 hours) and pharmacokinetic parameters of GSK2190915 will also be derived.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 65 years of age inclusive
* Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin ≤ 1.5x Upper limit of normal (ULN)
* Healthy as determined by a physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal . Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods. Those of child-bearing potential must agree to use one of the protocol contraception methods.
* Body mass index (BMI) within the range 18.5-29.0 kg/m2 (inclusive)
* Capable of giving written informed consent
* Current non-smokers who have not used tobacco products in the 6 month period preceding screening
* No significant abnormality on 12-lead electrocardiogram (ECG) at screening
* A 24 hour Holter ECG at screening that demonstrates no clinically significant abnormalities

Exclusion Criteria:

* A physician deems the subject unsuitable for the study
* A screening Holter ECG tracing that reveals clinically concerning arrhythmias
* A blood pressure that is persistently higher than 140/90 millimetres of mercury (mmHg) at screening.
* A mean heart rate outside the range 40-90 beats per minute (bpm) at screening.
* History or presence of any medically significant disease, or any disorder. In particular, a family history of QT prolongation, of early or sudden cardiac death or of early cardiovascular disease.
* A positive result for Hepatitis B or Hepatitis C within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities
* A positive pre-study drug/alcohol screen
* A positive test for Human Immunodeficiency Virus (HIV) antibody
* History of regular alcohol consumption within 6 months of the study
* The subject has participated in a clinical trial and has received an investigational product within 3 months of the first dosing day in the current study
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements from 14 days before screening until the follow-up visit unless permitted by the investigator
* History of sensitivity to any of the study medications
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 3 month period
* Pregnant females
* Lactating females
* Unwillingness or inability to follow the procedures outlined in the protocol
* Subject is mentally or legally incapacitated

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in QTcF interval at each timepoint on Day 5 (average of at least 3 12-lead Holter ECG replicates per time point) for 100mg GSK2190915 as compared with time-matched placebo | 5 days

SECONDARY OUTCOMES:
Change from baseline in QTcF interval at each timepoint on Day 5 (average of at least 3 12-lead Holter ECG replicates per time point) for 1000mg GSK2190915 as compared with time-matched placebo | 5 days
Change from baseline in QTcB interval at each timepoint on Day 5 (average of at least 3 12-lead Holter ECG replicates per time point) for 100mg and 1000mg GSK2190915 as compared with time-matched placebo | 5 days
Change from baseline in QTcF interval at each timepoint on Day 5 (average of at least 3 12-lead Holter ECG replicates per time point) for moxifloxacin as compared with time-matched placebo | 5 days
Plasma concentrations of GSK2190915 taken on Day 5 to derive pharmacokinetic parameters including Maximum observed concentration (Cmax), Time of occurrence of Cmax (tmax) and Area under the concentration-time curve over the dosing interval (AUC(0-τ)) | 5 days
Heart rate and ECG parameters taken on Day 1 and Day 5 compared with concentration of Plasma GSK2190915 to find relationship | 5 days
Maximal change from baseline on Day 5 for QTcF and QTcB | 5 days
Change from baseline at each timepoint on Day 5 for other cardiac electrophysiological parameters: QT, QRS, RR, PR and ventricular rate | 5 days
Assessment of safety and tolerability of GSK2190915 by 12-lead ECGs, vital signs, adverse events and clinical laboratory tests throughout treatment period | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom